CLINICAL TRIAL: NCT07345806
Title: Promoting Wellbeing and Personal Values: A Pilot Study on a Group-Based Program for Individuals With Special Needs and Their Caregivers
Brief Title: A Pilot Study on an ACT-Based Program for Individuals With Special Needs and Their Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Salvation Army, Hong Kong and Macau Command (Other)
Responsible Party: Principal Investigator, Amanda Kingsze CHEUNG, Research Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA250563
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Parenting Stress; Psychological Flexibility
Keywords: Acceptance and Commitment Therapy; Adults with SENs; Parents of Children with SENs
MeSH Terms: interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Acceptance and Commitment Therapy
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Acceptance and Commitment Therapy (ACT) is a well-established and evidence-based psychotherapy for individuals at different ages and with different clinical needs. The protocol used in the current study is adapted from an established local group intervention and tailored to families of individuals with special health care needs.

SUMMARY:
Parenting children with special health care needs can be stressful and weigh on the caregivers' mental health. For the individuals with special needs, the mismatch between their needs and the normative practice in the world around them can be frustrating and detrimental to their functioning. The demands and concerns to these families can be so real that it may not be sensible to examine the validity or helpfulness of the distressing thoughts or feelings but to promote psychological flexibility, which is a key to value-guided living. This pilot study explores the effects and feasibility of a group-based intervention for families of individuals with special health care needs.

ELIGIBILITY:
Inclusion Criteria:

* be at or older than 18 years old
* understand Cantonese
* read as well as write Chinese

Exclusion Criteria:

* with borderline or greater intellectual deficits
* weak language abilities
* severe conditions related to mental, emotional, and/or behavioral functioning

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Psychological Flexibility as Measured by the Multidimensional Psychological Flexibility Inventory | From baseline (T0) to two (T1), four (T2), and six (T3; post-intervention) weeks into treatment
  Score on psychological flexibility is the sum of scores across items
Change from Baseline in Psychological Inflexibility as Measured by the Multidimensional Psychological Flexibility Inventory | From baseline (T0) to two (T1), four (T2), and six (T3; post-intervention) weeks into treatment
  Score on psychological inflexibility is the sum of scores across items
Change from Baseline in Psychological Well-being as Measured by the 5-Item World Health Organization Well-being Index | From baseline (T0) to two (T1), four (T2), and six (T3; post-intervention) weeks into treatment
  Score on psychological well-being is the sum of scores across items
Change from Baseline in Parenting Stress as Measured by the Parenting Stress Scale | From baseline to six weeks into treatment
  Score on parenting stress is the sum of scores across items

SECONDARY OUTCOMES:
Change from Baseline in Child Externalizing as Measured by the Strengths and Difficulties Questionnaire | From baseline to six weeks into treatment (i.e., post-intervention)
  Score on externalizing is the sum of scores across items
Change from Baseline in Child Internalizing as Measured by the Strengths and Difficulties Questionnaire | From baseline to six weeks into treatment (i.e., post-intervention)
  Score on externalizing is the sum of scores across items
Participants' Satisfaction with the Intervention Program | Six-week into treatment (i.e., post-intervention)
  Eight items on a 5-point Likert scale are designed specifically for this study to assess participants' experience with the treatment program.
Participants' Personal Narratives on Their Experience with the Intervention Program | Within six weeks after completing the treatment
  Both open-ended text items and interviews are utilized to invite participants' sharing of their experiences throughout the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The Salvation Army SKY Family and Child Development Centre, Mong Kok, Hong Kong

IPD SHARING:
Plan to Share IPD: No